CLINICAL TRIAL: NCT04126629
Title: Association of Hypertensive Disorder of Pregnancy With Sleep-disordered Breathing.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Cooper Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 19-028EX
Record Dates: First submitted 2019-10-11; First posted 2019-10-15 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Hypertensive Disorder of Pregnancy; Sleep-disordered Breathing
Keywords: Hypertensive Disorder of Pregnancy; Sleep-disordered Breathing; HDP; SDB
MeSH Terms: conditions — Toxemia; Sleep Apnea Syndromes

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Normotensive Group: Subject will be allocated to the experimental group based on the clinical characteristics of their blood pressure. This will be the normotensive group. Every attempt will be made to stratify both groups equally between second and third trimesters.
- Hypertensive Group: Subject will be allocated to the experimental group based on the clinical characteristics of their blood pressure. This will be the hypertensive group.Every attempt will be made to stratify both groups equally between second and third trimesters.

SUMMARY:
This study aims to assess the prevalence of sleep disorder breathing in pregnant women with a singleton gestation who develop hypertensive disorder of pregnancy (HDP) compared to women without HDP, when matched for gestational age and body mass index.

DETAILED DESCRIPTION:
Sleeping disorder breathing is not only underdiagnosed in the general population, but more specifically in pregnant women. Some recent research has found an association between sleep disorder breathing and preeclampsia. Both conditions have shown to be associated with worse pregnancy outcomes. Therefore, more research is needed to find the strength of these associations. By gathering more information, this provides investigators with an opportunity to see if there is a way to slow the progression of complications in preeclampsia through the management of sleep-disordered breathing. Preeclampsia continues to be one of the top reasons for maternal mortality in the U.S. and this percentage continues to grow each year. Through the study, investigators hope to bring awareness of the comorbidity and how its similar pathogenesis can potential exacerbate complications in pregnant women.

ELIGIBILITY:
Inclusion Criteria:

* 1. Subject who is capable of consenting in English
* 2.Women with a diagnosis of a hypertensive disorder of pregnancy
* 3.Greater than 20 weeks pregnant
* 4.Singleton fetus
* 5.Inpatient

Exclusion Criteria:

* 1.With acute respiratory distress, including asthma
* 2.With micrognathia and other severe craniofacial abnormalities
* 3.Active heart failure
* 4.Sepsis
* 5.Subjects in labor.

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Pregnant women with a singleton gestation who are admitted to Cooper University Hospital that are greater than 20 weeks pregnant.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-01-22 (Estimated); Primary Completion 2020-09-01 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence of SDB in women with HDP compared to normotensive women. | 03/01/2019-03/01/2021

CONTACTS AND LOCATIONS:
Overall Officials: Meena Khandelwal, MD, Principal Investigator — Cooper Health System
Locations (1):
- Cooper University Hospital, Camden, New Jersey, United States

REFERENCES:
- [Background] Facco FL, Parker CB, Reddy UM, Silver RM, Koch MA, Louis JM, Basner RC, Chung JH, Nhan-Chang CL, Pien GW, Redline S, Grobman WA, Wing DA, Simhan HN, Haas DM, Mercer BM, Parry S, Mobley D, Hunter S, Saade GR, Schubert FP, Zee PC. Association Between Sleep-Disordered Breathing and Hypertensive Disorders of Pregnancy and Gestational Diabetes Mellitus. Obstet Gynecol. 2017 Jan;129(1):31-41. doi: 10.1097/AOG.0000000000001805. PMID 27926645
- [Background] Louis JM, Koch MA, Reddy UM, Silver RM, Parker CB, Facco FL, Redline S, Nhan-Chang CL, Chung JH, Pien GW, Basner RC, Grobman WA, Wing DA, Simhan HN, Haas DM, Mercer BM, Parry S, Mobley D, Carper B, Saade GR, Schubert FP, Zee PC. Predictors of sleep-disordered breathing in pregnancy. Am J Obstet Gynecol. 2018 May;218(5):521.e1-521.e12. doi: 10.1016/j.ajog.2018.01.031. Epub 2018 Feb 2. PMID 29523262
- [Background] Bourjeily G, Danilack VA, Bublitz MH, Lipkind H, Muri J, Caldwell D, Tong I, Rosene-Montella K. Obstructive sleep apnea in pregnancy is associated with adverse maternal outcomes: a national cohort. Sleep Med. 2017 Oct;38:50-57. doi: 10.1016/j.sleep.2017.06.035. Epub 2017 Jul 26. PMID 29031756